CLINICAL TRIAL: NCT07280650
Title: Feasibility and Acceptability of Earkick for Family Caregivers: Evaluation Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Noelle E Carlozzi, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00265379
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Caregivers
Keywords: Caregivers for adults with Traumatic Brain Injury (TBI); Caregivers for adults with dementia; Caregivers for adults with Huntington disease; Artificial intelligence (AI) mobile application; Chatbot; Surveys

STUDY DESIGN:
Intervention Model Description: The study will recruit approximately 20 care partners of individuals with TBI, 20 care partners of individuals with dementia, and 20 care partners of individuals with Huntington Disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Earkick app (Experimental)
  Interventions: Other: Earkick app

INTERVENTIONS:
Other: Earkick app — Participants will download the app with the study team's help and set it up. The participants will select topics of interest to focus on during the 8-week use of the Earkick app. Participants will choose one mental health related topic to focus on from weeks 1-4 and one physical health related topic to focus on from weeks 5-8. During these 4 week cycles the participants will be guided to engage with the app's "Chat" feature, which offers conversational support through interactions with the chatbot. Additionally, participants will complete surveys at baseline, the midpoint, and end of the 8-week intervention period. Participants will also complete a semi-structured interview to discuss their experience using the Earkick app.

SUMMARY:
This study evaluates the feasibility and acceptability of using the artificial intelligence (AI) chatbot mobile application (called Earkick) to support the well-being of informal care partners of individuals with traumatic brain injury (TBI), dementia, or Huntington disease (HD). Over an 8-week intervention period, up to 60 care partners will engage with the application (app), spending four weeks focusing on physical health and four weeks focusing on mental health. Participants will complete surveys at the midpoint and end of the intervention period. Participants will also complete a semi-structured interview to discuss participants experience using the Earkick app.

The study team hypothesizes that care partners will find the chatbot acceptable and feasible to use in daily life, and that there will be low attrition and high completion rates of the study.

ELIGIBILITY:
Inclusion Criteria (care partner)

* Age 18 years or older
* Able to independently provide informed consent
* Able to read, speak, and understand English
* Have an Apple (iOS) smartphone, tablet, or laptop, have access to the internet and text messages, and be willing to use these resources for the study, including downloading and using the AI chatbot app (Earkick)
* Be caring for and adult with a medically documented diagnosis of TBI, dementia or Huntington disease (HD)
* Provide emotional, physical, and/or financial support/assistance to the individual with the TBI, dementia, or HD, indicating a response per protocol
* Indicate high levels of caregiver burden, confirmed using the 12-item Zarit Burden questionnaire (scores must be ≥20)
* Willing to complete all study assessments for the duration of their study participation

Inclusion Criteria (care recipient):

* Age 18 years or older
* Have a medically documented diagnosis of TBI, dementia or Huntington disease as noted per protocol

Exclusion Criteria (care partner)

* Anyone not meeting inclusion criteria above
* Professional, paid caregivers
* Anyone at the discretion of the Principal investigator (PI) that would be a preclusion of safe or meaningful participation

Exclusion Criteria (care recipient):

* Anyone not meeting inclusion criteria
* Lives in a care facility (assisted living, nursing home) or is bedbound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability as measured by the Feasibility Questionnaire | 8 weeks (post intervention)
  Feasibility Questionnaire (items are scaled from 1 to 5 to indicate level of agreement, where "1" indicates "strong disagreement" and "5" indicates "strong agreement"). Feasibility and Acceptability as measured by ≥80% of participants indicating that care partners either "Agree" or "Strongly Agree" that the different study elements are feasible and acceptable.

SECONDARY OUTCOMES:
Attrition as measured by the percent of participants completing the study | Baseline to post intervention interview (approximately 8-12 weeks)
  The study team expects ≥80% of participants to complete the study.
Adherence as measured by the percentage of missing data over the course of the study | Baseline to 8 weeks
  Percent missing data of total expected data for each person and on average will also be calculated to characterize the feasibility of this approach (i.e., the study team expects ≥80% completion rates for the midpoint and end-of-study assessments).

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Carlozzi, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data collected during the trial, after de-identification, will be available for sharing with individuals in the scientific community, upon request, at the discretion of the Principal Investigator. The data will be available after the acceptance for publication of the main findings from the final dataset. The University of Michigan project manager will coordinate requests for data and maintain documentation for requests and distributions. An institutional data use agreement will be required before data is shared.
Time Frame: The data will be available after the acceptance for publication of the main findings from the final dataset.
Access Criteria: Data is available upon request to the project manager. Requests for data sharing should be emailed to PMR-CODALab@med.umich.edu